CLINICAL TRIAL: NCT04204213
Title: The 8 Section Brocade Tai Chi Therapy in Disease Management Program for Advanced Knee Osteoarthritis Patients: A Community - Based Care Approach
Brief Title: The 8 Section Brocade Tai Chi Therapy for Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Ho Ki Wai, Clinical Professional Consultant, Chinese University of Hong Kong
Other Study IDs: 3505.2715
Record Dates: First submitted 2019-12-15; First posted 2019-12-18 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Osteoarthritis, Knee; Tai Chi; Exercise Training
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Aquatic Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 8 Section Brocade Tai Chi Therapy: Subject participants with end stage osteoarthritis knee were enrolled into a customised multidisciplinary education program that consisted of one hour healthcare education seminars followed by another hour of 8 Section Brocade (Baduanjin) sitting Tai Chi classes for 4 consecutive weeks.
  Interventions: Behavioral: Tai Chi Exercise

INTERVENTIONS:
Behavioral: Tai Chi Exercise — 8 Section Brocade (Baduanjin) sitting Tai Chi classes + Healthcare Education seminars

SUMMARY:
Tai Chi exercises have increasingly grown in popularity among older adults in the past decades. It has been well studied to its efficacies in proportion with the management of elderly fall prevention and mineral-structured bone density enhancement. Nevertheless, existing study sources do little exemplified a quantifiable measures of effects in patients suffer from osteoarthritis of knees being impacted from a routine performance of Tai Chi.

DETAILED DESCRIPTION:
112 patients with end stage osteoarthritis knee had enrolled into a customised multidisciplinary education program that consisted of one hour healthcare education seminars followed by another hour of 8 Section Brocade (Baduanjin) sitting Tai Chi classes for 4 consecutive weeks. Followup measures were taken at baseline, 3 and 6 months post course commencement using the International Physical Activity Questionnaire (IPAQ), Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), SF-36v2 Health Survey and the Client Satisfaction Questionnaire (CSQ-8).

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed in symptomatic knee OA of Kellgren Lawrence (KL) grade 3 or 4, and have elected on list waiting for lower limb arthroplasty surgery
2. Aged 55 or above
3. Able to ambulate independently
4. Able to communicate in Cantonese

   Exclusion Criteria:
5. Previously underwent total knee replacement surgery
6. Diagnosed with other non-OA arthritide forms of the knees
7. Unable to complete all four sessions
8. Unable to complete all time-point measurements

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population with knee osteoarthritis.
Sampling Method: Non-Probability Sample
Enrollment: 112 (Actual)
Dates: Start 2015-01-31 (Actual); Primary Completion 2016-06-30 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Total physical activity metabolic equivalent of task (MET)-minutes per week | 6 Months
  The international Physical Activity Questionnaire-Short Form is designed to measure physical activity, and standardize measures of health-related physical activity behavior through 8 questions and divide patients into 3 activity groups. The health-enhancing physical activity level of category is for those people who either engaged in (1) ≥ 1500 MET-minutes on vigorous-intensity activity for at least three days, OR (2) at a combination of walking, moderate to vigorous intensity activities accumulative performance to ≥ 3000 MET-minutes per week. The Minimally Active level category is considered at the enrollment of (3) ≥ 20 mins vigorous activity for at least three days, OR (4) moderate-intensity activity or walking for ≥ 30 mins for at least five days, OR (5) any combination of walking, moderate/vigorous-intensity activities for at least 600 MET-minutes per week.

SECONDARY OUTCOMES:
Symptoms and Physical Functional Disability Scores | 6 Months
  The secondary outcome was shown by the symptoms and physical functional disability scores represented by the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) and the quality of life of participants represented by the self-rated questionnaire SF-36v2. WOMAC is a widely used standardized questionnaire to evaluate the condition of patients with osteoarthritis of the knee and hip, in three different domains for pain (score range 0 to 20), stiffness (0 to 8) and physical function (0 to 68).
Client Satisfactory Questionnaires Scores | 6 Months
  The Client Satisfactory Questionnaires (CSQ-8) is to assess the effectiveness of the customised programme and to collect feedback from a patient's point of view. Calculation on the 90 CSQ8 sampling sizes were made with the consideration on 95% confidence level, set with a 5% margin of error for the estimated confidence interval of 10. The CSQ-8 is a questionnaire that measures client satisfaction with services summing the individual item scores to produce a range of 8-32, with high scores indicating a greater satisfaction.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Orthopaedics & Traumatology, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Ho KK, Pong G, Poon QW, Kwok JY, Chau WW, Ong MT. A community-centric multi-disciplinary education program with the 8-section brocade Tai Chi therapy for patients with osteoarthritis of the knee - a pilot study. BMC Complement Med Ther. 2021 Dec 14;21(1):297. doi: 10.1186/s12906-021-03480-2. PMID 34906130